CLINICAL TRIAL: NCT04848935
Title: CURATE.AI Optimised Digital COgnitive Rehabilitation Therapy (COR-Tx) for Post Brain Radiotherapy Patients: CURATE.AI COR-Tx Mixed-methods Feasibility Clinical Trial
Brief Title: CURATE.AI COR-Tx Trial for Post Brain Radiotherapy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); The N.1 Institute for Health (N.1) (Other)
Responsible Party: Principal Investigator, Radiation Oncology, Principal Investigator, National University Hospital, Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020/00249
Record Dates: First submitted 2021-03-02; First posted 2021-04-19 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Cognitive Decline
Keywords: Oncology; Digital therapeutics; Cognitive evaluation; Digital diagnostic; Cognitive training; Phenotypic Personalised Medicine (PPM); Multi-Attribute Task Battery (MATB); Training intensity; Radiotherapy; CURATE.AI
MeSH Terms: conditions — Cognitive Dysfunction; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CURATE.AI (Experimental): A cognitive evaluation and a Digital Diagnostic (DD) session performed anytime before radiotherapy will serve as the baseline. After the radiotherapy treatment, which can last between 1 to 6.5 weeks, patients will have a variable recovery time (0 to 4 weeks). Subsequently, patients will be subject to a cognitive evaluation and a DD session, right before starting the Digital Intervention (DI) training. This training will comprise ten weeks of DI (three 10-15 minute sessions per week). Patients will complete cognitive evaluations and DD sessions at the end of DI, and 16 and 32 weeks after the end of DI.
  Interventions: Device: CURATE.AI

INTERVENTIONS:
Device: CURATE.AI — CURATE.AI will be utilised to provide personalised training intensity recommendations (low, medium or high) to the patients during the digital cognitive test battery DI session. The difficulty of each task will be modulated by CURATE.AI by adjusting the frequency of critical events that demand evaluation and/or response.

SUMMARY:
Cognitive deficit is common in patients who have undergone whole brain or partial brain radiotherapy. To counteract intellectual deterioration, the conventional strategies includes drug- based treatments such as donezepil and memantine, which have shown to only provide marginal improvement and, cognitive training regimens, both of which are usually administered at fixed dose/intensities often leading to sub-optimal responses. This study aims to address this clinically relevant problem by harnessing the CURATE.AI platform to identify N-of-1cognitive training profiles the can enhance learning trajectories through individualised calibration and training regimens. CURATE.AI is a phenotypic personalised medicine (PPM) platform that correlates a patient's phenotypic response (cognitive performance) to a certain input (training intensity) based exclusively on the patient's data. This PPM platform is independent of biological system or interventional agent and can be applied to any disorder treatment where dosing/intensity could be better personalised. CURATE.AI is expected to optimise/personalise cognitive training in post-brain radiotherapy patients by dynamically modulating the intensity of a digital cognitive test battery that measures executive processing, multitasking and perceptual learning tasks. In addition, this clinical feasibility trial aims to assess this cognitive test battery as a potential analogous or complementary diagnostic tool as compared to traditional cognitive evaluations performed by a clinician.

DETAILED DESCRIPTION:
Brain radiotherapy causes downstream cognitive deficits. Drug-based cognitive decline treatments show little improvement and side effects may reduce patient compliance. Regimens are usually administered at a fixed dose that doesn't incorporate high patient variability, leading to sub-optimal responses.

Effective cognitive training can improve cognitive performance. Artificial intelligence platforms show great potential for training personalisation. The CURATE.AI platform can be used to identify N-of-1 (single subject) training profiles that can be used to optimise learning trajectories through individualised calibration and training regimens, potentially leading to improved outcomes compared to standard static or adaptive training strategies. CURATE.AI uses only a subject's own performance data to identify the intensity needed for his/her best output. As the subject evolves during the course of intervention, the training intensities are dynamically modulated to maintain performance within a given range.

Here the investigators propose to test the feasibility of CURATE.AI, with a digital cognitive test battery as the interface, as an adaptive training platform for cognitive training addressed to improve brain cancer radiotherapy patients' cognitive performance. The acceptability, implementation and limited efficacy of the digital intervention (DI) will be explored. In addition, the investigators propose to test the feasibility of the digital cognitive test battery potential as a digital diagnostic (DD) tool as compared to traditional cognitive evaluations performed by a clinician. User experience and usability will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age >21 years.
* ECOG performance status 0 to 2.
* Patients with a neoplastic condition (benign or malignant) involving the brain or skull requiring radiotherapy (with or without chemotherapy).
* Patients with a life expectancy of at least 6 months.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Patients undergoing stereotactic radiosurgery (single fraction).
* Patients who are undergoing re-irradiation to the same area of the brain.
* Patients physically incapable of using computer tablet (either due to vision loss or dominant hand weakness)
* Patients who cannot understand spoken English language.
* Patients who are unable to give informed consent.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Patient acceptability of the digital cognitive test battery DI/DD obtained during a semi-structured interview | One visit 60 minutes (at the end of the 10 week intervention)
  Qualitative summary of patient acceptability of the digital cognitive test battery DI/DD
Patient adherence to the DI/DD | up to 12 months
  Percentage of completed DI/DD sessions
Patient attrition rate to the DI/DD | up to 12 months
  Percentage of patients that drop out of DI/DD
Percentage of CURATE.AI profiles successfully created and applied | up to 12 months
Timely delivery of DI/DD at indicated time points | up to 12 months
  Percentage of DI/DD sessions successfully delivered by study team at indicated time points
Digital intervention limited efficacy | up to 12 months
  Change in cognitive performance as measured by the standard of care cognitive evaluations pre-post digital intervention
Digital diagnostic limited efficacy | up to 12 months
  Correlation between standard of care cognitive evaluations scores and digital diagnostic scores

SECONDARY OUTCOMES:
1. Usability of the digital cognitive test battery DI/DD obtained during a semi-structured interview | One visit 60 minutes (at the end of the 10 week intervention)
  Qualitative summary of patient usability of the digital cognitive test battery DI/DD

CONTACTS AND LOCATIONS:
Overall Officials: Dr Balamurugan A Vellayappan, Principal Investigator — National University of Singapore
Locations (2):
- Singapore (2):
  - National University Hospital, Singapore
  - The N.1 Institute for Health (N.1), NUS, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kee, Theodore & Weiyan, Chee & Blasiak, Agata & Chong, Jordan & Chen, Jonna & Yeo, B.T. Thomas & Ho, Dean & Asplund, Christopher. (2019). Harnessing CURATE.AI as a Digital Therapeutics Platform by Identifying N-of-1 Learning Trajectory Profiles. Advanced Therapeutics. 2. 1900023. 10.1002/adtp.201900023.
- [Background] Zarrinpar A, Lee DK, Silva A, Datta N, Kee T, Eriksen C, Weigle K, Agopian V, Kaldas F, Farmer D, Wang SE, Busuttil R, Ho CM, Ho D. Individualizing liver transplant immunosuppression using a phenotypic personalized medicine platform. Sci Transl Med. 2016 Apr 6;8(333):333ra49. doi: 10.1126/scitranslmed.aac5954. PMID 27053773
- [Background] Pantuck AJ, Lee DK, Kee T, Wang P, Lakhotia S, Silverman MH, Mathis C, Drakaki A, Belldegrun AS, Ho CM, Ho D. Modulating BET bromodomain inhibitor ZEN-3694 and enzalutamide combination dosing in a metastatic prostate cancer patient using CURATE. AI, an artificial intelligence platform. Advanced Therapeutics. 2018 Oct;1(6):1800104.
- [Derived] Remus A, Tadeo X, Kai GNS, Blasiak A, Kee T, Vijayakumar S, Nguyen L, Raczkowska MN, Chai QY, Aliyah F, Rusalovski Y, Teo K, Yeo TT, Wong ALA, Chia D, Asplund CL, Ho D, Vellayappan BA. CURATE.AI COR-Tx platform as a digital therapy and digital diagnostic for cognitive function in patients with brain tumour postradiotherapy treatment: protocol for a prospective mixed-methods feasibility clinical trial. BMJ Open. 2023 Oct 24;13(10):e077219. doi: 10.1136/bmjopen-2023-077219. PMID 37879700